CLINICAL TRIAL: NCT06915857
Title: A Topical Betamethasone Versus Moisturizer in Preventing Radiation Dermatitis in Large-Breasted Patients Treated in the Prone Position: A Randomized Phase III Trial
Brief Title: Topical Betamethasone Versus Moisturizer in Preventing Radiation Dermatitis in Large-Breasted Patients Treated in the Prone Position
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Edward Chow, Co-Principal Investigator with Dr. Danny Vesprini [dvesprini] and Dr. Irene Karam [ikaram], Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Betamethasone RCT
Record Dates: First submitted 2025-03-17; First posted 2025-04-08 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Radiation Dermatitis
Keywords: Topical; Betamethasone; Prone position
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Intervention Model Description: Patients receiving whole or partial adjuvant breast radiation (RT) for invasive, in situ carcinoma of the breast or phyllodes who are at increased risk of developing moderate or severe radiation dermatitis (patients with large breasts [bra size 40 in and/or D cup or greater] and scheduled to be treated in the prone position receiving conventionally- (50Gy/25#), hypo-fractionated (40Gy/15#), or extreme hypo-fractionated (26Gy/5#) RT will be randomized in a 2:1 ratio to receive either 0.1% betamethasone cream or moisturizer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Betamethasone cream (Experimental): Patients randomized to the Betamethasone arm will receive the cream for the entire duration of their radiation treatment and will be worn up to 2 weeks after completion of radiotherapy. Patients randomized to this arm should not apply any standard of care treatments unless directed the treating radiation oncologist or nurse.
  Interventions: Device: Topical Betamethasone
- Standard of Care Arm (No Intervention): Patients randomized to the Standard of Care arm will be instructed to use the institutional standard of care skin treatments for the entire duration of their radiation treatment and up to 2 weeks after completion of radiotherapy.

INTERVENTIONS:
Device: Topical Betamethasone — Betamethasone a TC, reduces RD by promoting the synthesis of anti-inflammatory proteins while also preventing other inflammatory proteins from being synthesized
  Arms: Experimental Betamethasone cream

SUMMARY:
Radiotherapy (RT) is common in the treatment of breast cancer, however, 95% of breast cancer patients are at risk of developing acute and chronic skin toxicities known as radiation dermatitis (RD) which includes symptoms such as pruritus, edema, erythema, and moist desquamation (MD). Patients with a larger breast size are especially at risk of developing RD. The severity of RD can impact patient's quality of life (QOL) and their ability to complete treatment. Skin care guidelines for patients receiving RT vary and include barrier films and dressings, antibiotics, topical corticosteroids, and moisturizers. A study conducted at the Sunnybrook Odette Cancer Centre investigated the effectiveness of the prone treatment position during RT compared to the supine position. The results indicated that the prone position reduced the incidence of MD from 39.6% in supine to 26.9% in prone. However, 1 in 4 patients in the prone position still develop MD. Another study conducted at Sunnybrook Odette Cancer Centre found that Mepitel Film (MF), a barrier film, is more effective than the standard of care in preventing grade 2 or 3 RD, reducing the incidence of grade 2 or 3 RD from 45% to 15%. Despite its effectiveness, MF cannot be used for patients in the prone position and is costly. The topical corticosteroid betamethasone can prevent skin toxicity through its anti-inflammatory properties and is absorbed by the skin with minimal side effects. Betamethasone is cost-efficient and studies have found that it is effective in reducing the severity of RD in the supine position by half. Moreover, betamethasone can be applied in patients positioned in both prone and supine. The investigators hypothesize that adding betamethasone in large-breasted patients treated in prone during RT will further reduce RD.

This randomized control trial is the first of its kind to aim at investigating the effectiveness of betamethasone when compared with the standard of care in reducing the severity of RD in large-breasted patients being treated in the prone position during RT.

The investigators will enroll 276 breast cancer patients with band size ≥ 40 or ≥ D cup to be randomized to receive 0.1% betamethasone cream or the standard of care in a 2:1 ratio (alpha = 5% and power = 80% with the hypothesis that the addition of betamethasone to prone reduces the severity of RD from 30% to 15%). Upon enrolment, stratification factors will be recorded, and patients will be randomized into trial arms using procedures that balance stratification factors. All eligible patients will be stratified according to the following factors: patients receiving conventional RT (50Gy/25#) versus hypofractionated RT (40Gy/15#) versus extreme-hypofractionated RT (26Gy/5#), whole or partial breast radiation, patients with Fitzpatrick skin type VI versus patients with Fitzpatrick skin type I-V, patients receiving a planned boost versus patients without planned boost. The CRA will be responsible for collection of assessments and photos from patients. Patients will use the assigned cream daily during RT treatment and up until 2 weeks after RT. The primary endpoint of this study is acute grade 2 or 3 toxicities as defined by the Common Terminology Criteria for Adverse Events v5.0. Secondary endpoints will include patient- and clinician-reported outcomes as assessed by the Skin Symptom Assessment and the Radiation-Induced Skin Reaction Assessment Scale. Moreover, the investigators will also employ a QOL tool, the Skindex-16, and a Patient Satisfaction Questionnaire. Patients will complete assessments weekly during RT and 2 weeks post-RT in person, followed by 6 weekly assessments and a 3-month telephone follow-up post-RT. Clinicians will assess patients weekly during RT and at the 2-week follow-up appointment.

DETAILED DESCRIPTION:
Breast cancer is the most common female cancer in Canada. Breast cancer patients treated with a lumpectomy require adjuvant radiotherapy (RT) to achieve local control. Radiation dermatitis (RD) is a common radiation induced toxicity that affects up to 95% of all patients and can negatively impact quality of life (QOL). RD often presents as erythema, pruritus, and/or edema. In severe cases, skin breakage can occur resulting in moist desquamation (MD).

A randomized controlled trial (RCT) by De Langhe et al. (n=377) investigated factors that affect the development of breast RD. In patients with large breast size, those who were positioned in prone had less acute skin toxicity than those positioned in supine. Specifically, the rate of Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or higher events was 62.8% in supine and 43.7% in prone. A large confirmatory RCT was led at Sunnybrook Odette Cancer Centre treated with conventional and hypofractionated radiotherapy comparing supine and prone positions in women with large breast sizes (n=357). In this study, large breast size was classified with at least a cup size D or a band size 40 inches. The rates of MD decreased from 39.6% in the supine position to 26.9% for those in prone. While confirming the benefit of prone, this study demonstrates that one in four patients still develop MD. Additional interventions are therefore needed to further reduce RD in high-risk patients

Sunnybrook Odette Cancer Centre also performed a randomized controlled trial (RCT) (n=376) to study whether Mepitel Film (MF) was effective in preventing RD in patients with breast size at least a cup size C or a band size 36 in. MF is a silicone-based barrier film adhered to the skin to protect it during RT. Impressively, MF reduced rates of CTCAE grade 2 or 3 RD from 45.6% to 15.5% in patients treated in supine. However, patients with a large breast size did not tolerate MF well due poor film adherence and potential distortion of the breast contour. Therefore, the rates of RD in this group is not satisfactory. Furthermore, MF cannot be used for patients receiving RT in prone.

Topical corticosteroids (TCs) are another proven prophylactic intervention for RD which may be less resource-intensive and less expensive than MF, and can be applied in various treatment positions, such as in prone. TCs reduce RD through reducing inflammation in the skin and have been used for both the prevention and management of RD.

Mometasone furoate (MMF) is a TC that reduces inflammation by inducing the synthesis of proteins that inhibit phospholipase A2, thereby inhibiting the release of arachidonic acid from the cell membrane. A double blinded RCT by Miller et al. (n=166) investigated the effect of 0.1% MMF on acute skin toxicity. The incidence of CTCAE grade 2 or 3 RD was found to be 35.7% and 45.1% for MMF and placebo arms, respectively. Another double blinded RCT (n=124) investigated MMF's ability to reduce RD in post-mastectomy breast cancer patients. In this study, rates of CTCAE grade 2 or 3 RD were found to be 85.9% in the MMF arm and 96.7% in the standard arm. Rates of MD were 43.8% and 66.7% in the MMF and standard arms, respectively. A third double blinded RCT by Hindley et al. (n=114) found the rates of Radiation Therapy Oncology Group (RTOG) grade 2 or higher reactions to be 41.9% and 58.6% in the MMF arm and standard arm using an aqueous cream, respectively.

Betamethasone, another TC, reduces RD by promoting the synthesis of anti-inflammatory proteins while also preventing other inflammatory proteins from being synthesized. A double blinded RCT (n=102) led by Ulff et al. investigated the efficacy of using betamethasone and an emollient in reducing RD in comparison to two emollient creams used alone. They found an incidence of RTOG grade 3 reaction of 30.6% (n=15/49) in the emollient arms and 13.2% (n=7/53) in the betamethasone arm. In the second double blinded RCT done by Ulff et al. (n=202), betamethasone was used prophylactically in comparison with a moisturizer. It was found that only 8 participants using betamethasone (n=102) developed MD, and 71.0% and 31.4% developed RTOG grade 2 or 3 skin reactions using moisturizer and betamethasone, respectively. An open-label study done by Uysal et al. (n=50) compared the use of betamethasone cream to a moisturizer. In this study, no incidence of MD was found, and rates of 20.8% and 42.3% CTCAE grade 2 RD were observed using betamethasone and moisturizer, respectively.

Based on current literature, MMF reduced rates of grade 2 or 3 RD by 20-30%. In contrast, betamethasone reduced rates of grade 2 or 3 RD by around 50% in 3 RCTs. Notably, this near 50% reduction of RD was seen in both blinded studies and an open-label study. Therefore, it is feasible to perform an open-label RCT on the efficacy of topical betamethasone without significant bias. The investigators also performed a network meta-analysis of all RCTs that studied prophylactic TCs. This analysis showed that betamethasone is more efficacious in reducing the incidence of grade 2 or 3 RD compared to MMF (manuscript under preparation, results can be presented upon request from the PI). Additionally, there is data indicating that acute radiation dermatitis may disproportionately affect Black or African American patients.

The investigators will enroll 276 breast cancer patients with band size ≥ 40 or ≥ D cup to be randomized to receive 0.1% betamethasone cream or the standard of care in a 2:1 ratio (alpha = 5% and power = 80% with the hypothesis that the addition of betamethasone to prone reduces the severity of RD from 30% to 15%). Upon enrolment, stratification factors will be recorded, and patients will be randomized into trial arms using procedures that balance stratification factors. All eligible patients will be stratified according to the following factors: patients receiving conventional RT (50Gy/25#) versus hypofractionated RT (40Gy/15#) versus extreme-hypofractionated RT (26Gy/5#), whole or partial breast radiation, patients with Fitzpatrick skin type VI versus patients with Fitzpatrick skin type I-V, patients receiving a planned boost versus patients without planned boost.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Female.
* Histological confirmation of breast malignancy (invasive or in situ carcinoma) or phyllodes.
* Patients with large breasts [bra size 40 in and/or D cup or greater] and have undergone breast-conserving surgery.
* Patients are scheduled to receive conventionally- (50Gy/25#), hypo-fractionated (40Gy/15#), or extreme hypo-fractionated (26Gy/5#) photon-based radiation to whole or partial breast in prone position.
* Patients treated with or without the addition of a boost.
* Patient speaks English or can be aided by a translator.

Exclusion Criteria:

* Patients planning brachytherapy within the treatment field, and patients scheduled to receive bilateral radiation.
* Prior RT to any portion of the planned treatment site.
* Active rash or pre-existing dermatitis within the treatment field.
* Concomitant cytotoxic chemotherapy.
* Unable to tolerate RT in prone.
* Treatment involves use of tissue equivalent bolus.
* Known sensitivity or allergy to betamethasone.
* Known pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-09-06 (Estimated); Study Completion 2026-12-06 (Estimated)

PRIMARY OUTCOMES:
Acute grade 2 or 3 toxicities as defined by the CTCAE v5.0 assessed by HCP | Within 3 months following radiation
  The efficacy of the steroid, 0.1% betamethasone cream, versus the institutional standard of care in reducing acute grade 2 or 3 toxicities in patients undergoing whole or partial breast RT based on the Common Terminology Criteria for Adverse Events (CTCAE) v.5.0 assessed by HCPs, comparing changes in the treated versus non-treated breast or chest wall from baseline to weekly during radiation treatment and 2 weeks post radiation treatment.
  CTCAE Dermatitis Grade (higher scores mean worse outcome): 0 No symptoms, 1 Faint erythema or dry desquamation, 2 Moderate to brisk erythema; patchy moist desquamation, mostly confined to skin fold and creases; moderate edema, 3 Moist desquamation in areas other than skin folds and creases; bleeding induced by minor trauma or abrasion, 4 Life-threatening consequences; skin necrosis or ulceration of full thickness dermis; spontaneous bleeding from involved site; skin graft indicated, 5 Death

SECONDARY OUTCOMES:
Patient-reported skin-related symptoms using the Skin Symptom Assessment (SSA) | Within 3 months following radiation
  Patient assessed Skin Symptom Assessment (SSA) scores obtained at baseline compared to scores obtained once weekly during RT, 14 days (+/- 4 days) post-RT in-person, during weeks 1 and 3-6 post-RT on telephone, and 3 months post-RT. The SSA measures pruritus (itchiness), pain or soreness, blistering or peeling, erythema (redness), pigmentation (discolouration/darkness), edema (swelling), and trouble fitting brassieres using the scales: none, mild, moderate, severe.
Clinician-assessed skin-related symptoms using the Skin Symptom Assessment (SSA) | Within 3 months following radiation
  RD severity is based on clinician-assessed Skin Symptom Assessment (SSA) scores obtained at baseline compared to scores obtained once weekly during RT, and 14 days (± 4 days) post-RT in-person. The SSA measures pruritus (itchiness), pain or soreness, blistering or peeling, erythema (redness), pigmentation (discolouration/darkness), edema (swelling), and trouble fitting brassieres using the scales: none, mild, moderate, severe.
Photographs of treated and non-treated breast/chest wall for blind and unbiased assessment of the skin by HCPs | Within 3 months following radiation
  Photographs of the patient's treated and non-treated breast/chest wall will be taken and used for blind and unbiased assessment of the skin by a group of health care professionals. These results can be compared to in person assessments as scaled on the CTCAE, RISRAS, and the SSA. Patient photos will be taken at baseline when the patient is first recruited, the last treatment day of radiation (3-5 weeks after the first day of radiation depending on radiation dose/fractionation) and at 2 weeks follow up after the end of radiation.
Radiation-Induced Skin Reaction Assessment Scale (RISRAS) assessed by patient | Within 3 months following radiation
  RD severity is based on patient-assessed Radiation-induced Skin Reaction Assessment Scale (RISRAS) scores obtained at baseline compared to scores obtained at the patient's final review appointment, 14 days (± 4 days) post-RT in-person, and 3 months post-RT. Patient-assessed RISRAS scores range from 0-3, with higher scores meaning worse outcome.
Radiation-Induced Skin Reaction Assessment Scale (RISRAS) assessed by HCP | Within 3 months following radiation
  RD severity is based on HCP-assessed Radiation-induced Skin Reaction Assessment Scale (RISRAS) scores obtained at baseline compared to scores obtained at the patient's final review appointment, 14 days (± 4 days) post-RT in-person, and 3 months post-RT. Provider-assessed RISRAS scores obtained at baseline are compared to scores obtained at the patient's final review appointment, 14 days (± 4 days) post-RT in-person. Provider-assessed RISRAS scores range from 0-4, with higher scores meaning worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Edward LW Chow, MBBS, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No